CLINICAL TRIAL: NCT06709586
Title: Thermal Ablation Versus Parathyroidectomy for Secondary Hyperparathyroidism: a Multicenter Study
Brief Title: Thermal Ablation Versus Parathyroidectomy for Secondary Hyperparathyroidism
Status: Not yet recruiting | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Ping Liang, Professor, Chinese PLA General Hospital
Other Study IDs: S2024-11-10
Record Dates: First submitted 2024-11-10; First posted 2024-11-29 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-06

CONDITIONS: Achievement Rate; Efficacy and Safety; PTH; Calcium; Clinical Symptoms
MeSH Terms: interventions — Transurethral Resection of Prostate; Parathyroidectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Therma ablation
  Interventions: Procedure: Thermal ablation
- Parathyroidectomy
  Interventions: Procedure: parathyroidectomy

INTERVENTIONS:
Procedure: Thermal ablation — Thermal ablation is a treatment for secondary hyperparathyroidism. There are radiofrequency ablation (RFA) and microwave ablation (MWA). For RFA, an electrode needle is inserted into the parathyroid under imaging guidance. High - frequency current heats the tissue to cause necrosis. MWA uses electromagnetic waves to generate heat by friction. Before ablation, imaging and lab tests are done for evaluation. During the process, precise positioning and real - time monitoring are key. After that, patients are observed for bleeding, swelling and other symptoms, and tests are repeated to assess the effect.
  Groups: Therma ablation
Procedure: parathyroidectomy — Parathyroidectomy for secondary hyperparathyroidism is a common approach. The surgeon first makes an incision in the neck area under general or local anesthesia. Then, the enlarged parathyroid glands are carefully identified and dissected. Precise surgical skills are required to avoid damaging nearby structures such as the recurrent laryngeal nerve and blood vessels. After the removal of the abnormal parathyroid tissue, the wound is closed.
  Groups: Parathyroidectomy

SUMMARY:
Secondary hyperparathyroidism (SHPT), which is frequently associated with chronic kidney disease, leads to problems such as bone pain, fractures, and cardiovascular issues, thereby affecting patients' quality of life. This clinical trial is designed to compare the efficacy of thermal ablation and surgical treatment for SHPT. Parameters including parathyroid hormone levels, serum calcium and phosphorus levels, SHPT-related symptoms (for example, bone pain, muscle weakness), and complication occurrence will be monitored. The advantages involve enabling better treatment decisions for patients, enhancing patients' quality of life, and alleviating the burden on families, in addition to augmenting the clinical knowledge of healthcare providers. However, both treatments carry risks. Thermal ablation may have problems like incomplete ablation, local tissue damage, and blood parameter changes. Surgical risks comprise bleeding, infection, adjacent tissue damage (such as the recurrent laryngeal nerve), and hypoparathyroidism. The investigators will strive to minimize these risks. This trial is of great significance for SHPT treatment, and the investigators welcome participants to contribute to the advancement of medical science in this area.

ELIGIBILITY:
Inclusion Criteria:

* persistent serum iPTH (intact parathyroid hormone) levels > 800 pg/mL；
* resistance to calcimimetics, vitamin D, and its analogs, with ineffective conventional internal medicine comprehensive treatment；
* severe bone pain, osteoporosis, muscle pain, ectopic soft tissue calcification, or other factors affecting quality of life；
* imaging examinations indicating the presence of at least one enlarged parathyroid gland

Exclusion Criteria:

* severe bleeding tendency or coagulation disorders, severe cardiopulmonary abnormalities, and abnormal vital signs such as severe hypertension, arrhythmias, and anemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients must have a confirmed diagnosis of secondary hyperparathyroidism based on clinical symptoms (such as bone pain, fractures, pruritus), biochemical parameters (elevated parathyroid hormone, abnormal calcium, phosphorus, and alkaline phosphatase levels), and relevant medical history (especially those with underlying chronic kidney disease or other relevant disorders). All patients must provide written informed consent after a detailed discussion of the study purpose, procedures, potential risks, and benefits of both treatment options by the research team.
Sampling Method: Non-Probability Sample
Enrollment: 612 (Estimated)
Dates: Start 2024-11-26 (Estimated); Primary Completion 2028-11-26 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Achievement rate of target PTH value | 6 months after surgery or ablation
Symptom remission rate | 1 year after treatment
  The symptom remission rate refers to the proportion of the number of patients whose symptoms have been alleviated to the total number of patients treated in the treatment of primary hyperparathyroidism, either by surgery or ablation.

SECONDARY OUTCOMES:
complication rate | within 30 days after surgery or ablation
  The incidence rate of complications refers to the proportion of patients who experience complications after a surgical procedure within a certain period.
Normalization Probability of Serum Calcium and Phosphorus after Ablation or Surgery | 6 months post-treatment
  The probability of normal serum calcium and serum phosphorus levels after ablation or surgical treatment for primary hyperparathyroidism is defined as the proportion of patients in whom the levels of blood calcium and blood phosphorus return to the normal physiological range among all the patients who have received either ablation or surgical procedures for this condition.
Bone mineral density change | 2 years
  Bone mineral density change after treatment is defined as the alteration in bone density measured by DEXA in patients with primary hyperparathyroidism after surgery or ablation.
Assessment of Changes in Bone Metabolism Markers Including BALP, PINP, and ALP for Treating Primary Hyperparathyroidism by Surgery and Ablation | 1 year
  Changes in Bone Metabolism Markers will be evaluated by measuring specific biochemical parameters. These include serum levels of bone-specific alkaline phosphatase (BALP), which is a biomarker reflecting osteoblast activity. Another important marker is N-terminal propeptide of type I collagen (PINP), which is involved in collagen synthesis and provides insights into bone formation. ALP is a well-known enzyme related to bone metabolism and its elevation can be indicative of increased osteoblastic activity. The levels of these markers will be determined using enzyme-linked immunosorbent assay (ELISA) kits, which are highly sensitive and specific laboratory assays.
All - cause mortality rate | 2 years

OTHER OUTCOMES:
Cosmetology Scoring（Scar Cosmesis Assessment and Rating Scale） | at 3 months, 6 months, and 1 year post-procedure
  The Scar Cosmesis Assessment and Rating Scale (SCAR) will be utilized to evaluate the cosmetic outcome following surgical or ablation treatment for primary hyperparathyroidism. The observer part of the SCAR assesses six aspects: scar spread, erythema, pigmentation abnormality, surgical marks or suture tracks, hypertrophy/atrophy, and overall impression. The patient part includes two simple questions about patient satisfaction with the scar and the degree of itching. The scale has a minimum value of 0, representing the least severe scar with the best cosmetic appearance, and a maximum value of 15, signifying the most severe scar with the poorest cosmetic result. Higher scores on this scale indicate a worse cosmetic outcome.
Readmission Rate within 30 Days | within 30 days after surgery or ablation
Evaluation of the Learning Curve for Surgical and Ablation Procedures in Treating Primary Hyperparathyroidism: Incorporating Key Performance Indicators and Patient Cure Outcomes | through study completion, an average of 2 year
  The learning curve for surgical or ablation procedures will be evaluated by tracking and analyzing key performance indicators, with patient cure outcomes also taken into account. These indicators encompass the time taken from the start of the procedure until its completion (operation time). Additionally, the rate of occurrence of immediate and short-term post-operative complications (like bleeding, nerve injury) is considered. Patient cure status, such as complete remission of related symptoms, normalization of relevant physiological indicators, and long-term disease-free survival, will be meticulously assessed to comprehensively evaluate the effectiveness and learning the effectiveness and learning curve of these procedures.

IPD SHARING:
Plan to Share IPD: No